CLINICAL TRIAL: NCT02594059
Title: Assessment of Peripheral Endothelial Function in Idiopathic Pulmonary Fibrosis
Acronym: Endoth-FPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/56
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Fibrosis
Keywords: endothelial function, idiopathic pulmonary fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary idiopathic fibrosis (Experimental): Patients with pulmonary idiopathic fibrosis according to ATS/ERS 2011's criteria
  Interventions: Other: endothelial function

INTERVENTIONS:
Other: endothelial function — measure of reactive hyperemia-peripheral artery tone index

SUMMARY:
The aim of the study is to assess the peripheral endothelial function in adult patients with idiopathic pulmonary fibrosis (IPF) and the relationship between the peripheral endothelial function and the severity of the IPF.

DETAILED DESCRIPTION:
The primary criteria is the peripheral endothelial function that will be assessed by the measure of flow-mediated dilation (reactive hyperemia-peripheral artery tone index). The pulmonary function will be assessed by the measures of the forced expiratory volume at one second (FEV1), the forced vital capacity (FVC) and the total lung capacity (TLC) and the diffusing capacity of the lung for carbon monoxide (DLCO). The dyspnea will be assessed with the New York Heart Association (NYHA) score. The exercise capacity will be assessed by the 6-min walk test. Pulmonary arterial pressure will be recorded through cardiac echography or catheterization.

ELIGIBILITY:
Inclusion Criteria:

* IPF according to ATS/ERS 2011's criteria
* Stable IPF (no reduction of FVC or DLCO of more than 10% and 15% respectively)

Exclusion Criteria:

* Patients with a significant disease other than IPF. A significant disease is defined as a disease which, in the opinion of the investigator, may influence the results of the trial.
* Pregnant or nursing women.
* Non-pulmonary fibrosis
* treatment by pulmonary vasodilators that cannot be stopped for 24 hours for the assessment of endothelial function

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
measure of reactive hyperemia-peripheral artery tone index | day 1

SECONDARY OUTCOMES:
endothelial function | 1, 2 and 3 years
  measure of reactive hyperemia-peripheral artery tone index
measure of reactive hyperemia-peripheral artery tone index | 3 years
  measure of reactive hyperemia-peripheral artery tone index at IPF exacerbation or PAHT's occurence

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Europeen Georges Pompidou, dpt of pneumology, Paris
  - Hopital Foch, Suresnes